CLINICAL TRIAL: NCT05903300
Title: Validation of the Polish Version of the Musculoskeletal Pain Intensity and Interference Questionnaire for Musicians (MPIIQM-P)
Brief Title: Validation of the Polish Version of the MPIIQM Questionnaire for Musicians
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Anna Cygańska (Other)
Responsible Party: Sponsor-Investigator, Anna Cygańska, Principal Investigator, PhD in physical culture science, Józef Piłsudski University of Physical Education
Organization: Józef Piłsudski University of Physical Education (Other)
Other Study IDs: SKE 01-01/2023
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Musculoskeletal Pain; Questionnaire
Keywords: Occupational Diseases; Musculoskeletal Pain; Questionnaires; Validation Studies; Pain Measurement
MeSH Terms: conditions — Musculoskeletal Pain; Occupational Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Professional orchestra musicians: The study group consists of adult, professionally active people (women and men) who are professional orchestra musicians. The mother tongue of the respondents must be Polish.
  Interventions: Other: Surveys and Questionnaires

INTERVENTIONS:
Other: Surveys and Questionnaires — The intervention consists of completing the MIPIM-P, QuickDash, and Brief Pain Inventory questionnaires.

SUMMARY:
The aim of this study, originally named "Cross-Cultural Adaptation and Validation of the Musculoskeletal Pain Intensity and Interference Questionnaire for Musicians of the Polish Population (MPIIQM-P)" is the enlargement of validation of the Polish questionnaire.

DETAILED DESCRIPTION:
The aim is to determine the following psychometric properties: convergent and divergent validity, two-time reliability analysis, and exploratory factor analysis according to the recommended number of subjects of ≥45 subjects. In addition, the aim of the study is to assess the psychometric properties of the MPIIQM-P questionnaire in the online version and to compare these results with the results for the paper version obtained by Cygańska et al., 2021.

ELIGIBILITY:
Inclusion Criteria:

* permanent musician in an orchestra
* Polish as a native language

Exclusion Criteria:

• freelance musician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group consists of adult, professionally active people (women and men) who are professional orchestra musicians. The mother tongue of the respondents must be Polish.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-10-28 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity MPIQIM | Baseline and change between baseline and after few (3/4) days
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P); The pain intensity score can be defined as the sum of the four pain intensity items (0-40, the higher the score, the greater the pain intensity) or the mean of pain intensity score (0-10, the higher the score, the greater the pain intensity).
Pain Intensity BPI | Baseline and change between baseline and after few (3/4) days
  In Brief Pain Inventory, subjects rates their pain intensity on a numeric rating scale from 0 to 10, the higher the score, the greater the pain intensity. The pain intensity score can be defined as the sum of the four pain intensity items (0-40, the higher the score, the greater the pain intensity). In the inventory, a score of 1-4 is defined as mild pain, a score of 5-6 as moderate pain, and a score of 7-10 as severe pain.
Pain Interference MPIQIM | Baseline
  The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians of the Polish Population (MPIIQM-P); The pain interference score can be defined as the sum of the four pain interference items (0-50, the higher the score, the greater the pain interference) or the mean of pain interference score (0-10, the higher the score, the greater the pain interference).
Pain Interference BPI | Baseline
  In Brief Pain Inventory, subjects rate their pain interference on a numeric rating scale from 0 to 10, the higher the score, the greater the pain interference. The pain interference score can be defined as the sum of the four pain interference items (0-70, the higher the score, the greater the pain intensity) or the mean of the pain interference score (0-10, the higher the score, the greater the pain interference).
Pain Interference | Baseline
  In Quick Dash Questionaire, subjects rate their pain interference on a numeric rating scale from 0 to 5, the higher the score, the greater the pain interference. The pain interference score can be defined as the sum of the selected answers, divided by 4 (i.e. number of questions), subtracting 1, and multiply by 25.

CONTACTS AND LOCATIONS:
Overall Officials: Anna K. Cygańska, Cygańska, Principal Investigator — Józef Piłsudski University of Physical Education in Warsaw
Locations (1):
- Józef Piłsudski University of Physical Education in Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No